CLINICAL TRIAL: NCT00022334
Title: A Phase I/II Trial Testing Immunization With Dendritic Cells Pulsed With Four AFP Peptides in Patients With Hepatocellular Carcinoma
Brief Title: Vaccine Therapy in Treating Patients With Liver Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068806; UCLA-0001026; NCI-G01-1997
Record Dates: First submitted 2001-08-10; First posted 2003-01-27 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2012-07

CONDITIONS: Liver Cancer
Keywords: localized resectable adult primary liver cancer; localized unresectable adult primary liver cancer; advanced adult primary liver cancer; recurrent adult primary liver cancer; adult primary hepatocellular carcinoma
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): See intervention description.
  Interventions: Biological: AFP

INTERVENTIONS:
Biological: AFP — Increasing doses of AFP will be given to groups of 3 intradermally. Subjects will receive 3 biweekly vaccinations. At least 2 patients at a given dose must have received their complete 3 vaccination schedule with a 30 day observation period after the last vaccination before a higher dose is initiated.
  Other Names: AFP peptide-pulsed autologous DC

SUMMARY:
RATIONALE: Vaccines made from a person's white blood cells mixed with tumor proteins may make the body build an immune response to kill tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of vaccine therapy in treating patients who have liver cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of alpha-fetoprotein peptide-pulsed autologous dendritic cells in HLA-A*0201-positive patients with hepatocellular carcinoma.
* Determine the safety and toxicity of this regimen in these patients.
* Determine the immunological effects of this regimen in these patients.
* Determine the progression-free survival and clinical responses in patients treated with this regimen.

OUTLINE: This is a dose-escalation study.

Patients receive alpha-fetoprotein peptide-pulsed autologous dendritic cells intradermally on day 1. Treatment repeats every 2 weeks for a total of 3 doses in the absence of unacceptable toxicity.

Cohorts of 3-12 patients receive escalating doses of vaccine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 or 2 of 12 patients experience dose-limiting toxicity.

Patients are followed at weeks 1, 4, and 12 and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 12-18 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* HLA-A*0201 positive adults over the age of 18.
* Have HCC with a serum AFP determination >30ng/ml.
* Both male and female patients may be enrolled.
* Karnofsky Performance Status greater than or equal to 70 percent.
* No previous evidence of class 3 or greater New York Heart Association cardiac insufficiency or coronary artery disease.
* No previous evidence of opportunistic infection.
* Adequate baseline hematological function as assessed by the following laboratory values with 30 days prior to study entry:

  1. Hemoglobin >9.0g/dl
  2. Platelets >50000/mm3
  3. Absolute Neutrophil Count >1,000/mm3
* Child-Pugh Class A or B for chronic liver disease.
* Ability to give informed consent.

Exclusion Criteria:

* Any congenital or acquired condition leading to inability to generate an immune response, including concomitant immune suppressive therapy.
* Concomitant steroid therapy or chemotherapy, or any of these other treatments < 30 days before the first vaccination.
* Females of child-bearing potential must have negative serum beta-HCG pregnancy test (within Day -14 to Day 0).
* Acute infection: any acute viral, bacterial, or fungal infection, which requires specific therapy. Acute therapy must have been completed within 14 days prior to study treatment.
* HIV-infected patients.
* Patients with any underlying conditions which would contraindicate therapy with study treatment.
* Patients with organ allografts.
* O2 sat <91% on room air; dyspnea at rest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2001-01; Primary Completion 2004-12 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity and maximum tolerable dose. | 1 year

SECONDARY OUTCOMES:
Generation of AFP specific immunity. | 3 years
Progression-free survival. | 3 years
clinical response in patients with measurable disease. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: James S. Economou, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States